CLINICAL TRIAL: NCT03363100
Title: Diabetes Coaching Program for Medicare Advantage Members With Type 2 Diabetes - Impact on A1c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidation Health (Industry)
Collaborators: Humana Co.Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EH-006
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Digital health Partnership program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Digital health Partnership program — The program pairs patients with their own certified diabetes educator coach who will guide the patient through a personalized program that leverages a proven educational curriculum combined with proven patient engagement methods.
  Arms: Intervention

SUMMARY:
The Diabetes Coaching Program for Medicare Advantage Members with Type 2 Diabetes - Impact on A1c trial is a 26-week long, prospective, intent-to-treat, 2-arm randomized controlled trial that aims to evaluate the impact of the Digital Health Partnership on A1c levels for individuals with uncontrolled Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Humana Medicare Advantage member
* Type 2 diabetes diagnosis
* HbA1c levels ≥ 8.0% verified by lab test

Exclusion Criteria:

* Has any of the following conditions: cancer, chronic heart failure, chronic obstructive pulmonary disease, respiratory failure, chronic kidney disease, end stage renal disease, peripheral vascular disease
* Not fluent in English
* Humana membership is part of a Full or Global risk arrangement
* Enrolled in Humana at Home Care Management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-02-23 (Actual)

PRIMARY OUTCOMES:
A1c | Baseline and 6 months
  Change in A1c from study baseline to study end for participants

CONTACTS AND LOCATIONS:
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No